CLINICAL TRIAL: NCT01821079
Title: A Phase 1, Single-Dose, Open-Label, Crossover Study To Assess The Relative Bioavailability Of Powder-In-Capsule And A Tablet Formulation Of Pf-05175157 And The Effect Of Food On The Pharmacokinetics Of The Tablet Formulation In Healthy Volunteers
Brief Title: A Healthy Volunteer Study To Assess Relative Bioavailability Of Powder-In-Capsule And A Tablet Formulation And The Effect Of Food On The Pharmacokinetics Of The Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1731014
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: Single dose; Relative Bioavailability; Food effect; Healthy subjects; Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-05175157 PIC in fed state (Experimental): 200 mg single dose of PF-05175157 administered as PIC in the fed state (following a standard high fat meal).
  Interventions: Drug: PF-05175157
- PF-05175157 tablet in fed state (Experimental): 200 mg single dose of PF-05175157 administered as tablet formulation in the fed state (following a standard high fat meal).
  Interventions: Drug: PF-05175157
- PF-05175157 tablet in fed state (repeat) (Experimental): 200 mg single dose of PF-05175157 administered as tablet formulation in the fed state (following a standard high fat meal).
  Interventions: Drug: PF-05175157
- PF-05175157 tablet in fasted state (Experimental): 200 mg single dose of PF-05175157 administered as tablet formulation in the fasted state (following at least a 10 hour fast).
  Interventions: Drug: PF-05175157

INTERVENTIONS:
Drug: PF-05175157 — Single 200 mg dose of PF-05175157 administered as powder in capsule (2x100 mg)
  Arms: PF-05175157 PIC in fed state
Drug: PF-05175157 — Single 200 mg dose of PF-05175157 administered as tablet formulation (2x100 mg)
  Arms: PF-05175157 tablet in fed state
Drug: PF-05175157 — Single 200 mg dose of PF-05175157 administered as tablet formulation (2x100 mg)
  Arms: PF-05175157 tablet in fed state (repeat)
Drug: PF-05175157 — Single 200 mg dose of PF-05175157 administered as tablet formulation (2x100 mg)
  Arms: PF-05175157 tablet in fasted state

SUMMARY:
The purpose of this study in healthy volunteers is to assess the relative bioavailability of PF-05175157 as powder-in-capsule and a tablet formulation and the effect of food on the pharmacokinetics of the tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive
* Women must be of non childbearing potential
* Body Mass Index (BMI) of 25 to 35 kg/m2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* Active ocular disease including infection, glaucoma, seasonal allergies, dry eye symptoms, optic nerve disease or retinal disease.
* History of habitual smoking in the past 5 years or history or evidence of habitual use of other (non smoked) tobacco or nicotine-containing products within 3 months of Screening or positive cotinine test at Screening or Day 0

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0 to 72 H after dose
Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf) | 0 to 72 H after dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0 to 72 H after dose
Time at which maximum plasma concentration is observed (Tmax) | 0 to 72 H after dose
Plasma Decay Half-Life (t1/2) | 0 to 72 H after dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1731014&StudyName=A%20Healthy%20Volunteer%20Study%20To%20Assess%20Relative%20Bioavailability%20Of%20Powder-In-Capsule%20And%20A%20Tablet%20Formulation%20And%20The%20Effect%20Of%20Food%20On%20T